CLINICAL TRIAL: NCT00845546
Title: Comparative, Randomized, Single-Dose, Fully Replicated, 4-Way Crossover Bioavailability Study of Ranbaxy and Schering (Claritin_D® 24 Hour) 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets, in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Loratadine / Pseudoephedrine Sulfate 10/ 240 mg Extended-Release Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA01112
Record Dates: First submitted 2009-01-08; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Bioequivalence 10 mg Loratadine 240 mg Pseudoephedrine Sulfate Extended Release Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets of Ranbaxy
  Interventions: Drug: 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets
- 2 (Active Comparator): (Claritin_D® 24 hour) 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets
  Interventions: Drug: 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets

INTERVENTIONS:
Drug: 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and Schering (Claritin-D® 24 hour) 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets, in a fully replicated design, under fed conditions.

DETAILED DESCRIPTION:
The study was conducted as an open-label, randomized, Single-Dose, Fully replicated, 4-way Crossover Study to compare the single-dose relative bioavailability of Ranbaxy and Schering (Claritin_D® 24 hour) 10 mg Loratadine/240 mg Pseudoephedrine Sulfate Extended-Release Tablets, in Healthy adult Volunteers Under Fed Conditions In each period, subjects were housed from the evenings before the dosing until after the 36 hour blood draw and were to return for subsequent blood draws at 48, 72, 96 and 120 hours post dose. Single oral 10 mg Loratadine/ 240 mg Pseudoephedrine Sulfate doses were separated by a washout period of 21 days.

A total of 40 subjects and 1 alternate (34 males and 7 females) were included in this study, of which 37 (32 males and 5 females) finished the study according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers, 18-45 years of agestart of the study.
* Other birth control methods may be deemed acceptable
* Postmenopausal women with amenorrhea for at least 2 years will be eligible
* Voluntarily consent to participate in the study

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* In addition, history or presence of:

  * alcoholism or drug abuse within the past year
  * hypersensitivity or idiosyncratic reaction to Loratadine or any other H1-receptor antagonist
  * hypersensitivity or idiosyncratic reaction to Pseudoephedrine or any other sympathomimetic amines
* Glaucoma or hypermetropia
* Subjects receiving a monoamine oxidase (MAO) inhibitor or within 14 days of stopping use of an MAO inhibitor, or any sympathomimetic amines
* Subjects who have used any drugs or other substances known to be strong inhibitors of CYP (cytochrome P450) enzymes within 10 days of study start
* Subjects who have used any drugs or other substances known to be strong inducers of CYP (cytochrome P450) enzymes within 28 days of study start
* Female subjects who are pregnant or lactating
* Subjects who have been on an abnormal diet (for whatever reason) during the 28 days prior to the first dose
* Subjects who, through completion of the study, would have donated in excess of:

  * 500 mL of blood in 14 days
  * 500-750 mL of blood in 14 days (unless approved by the principal Investigator)
  * 1000 mL of blood in 90 days
  * 1250 mL of blood in 120 days
  * 1500 mL of blood in 180 days
  * 2000 mL of blood in 270 days
  * 2500 mL of blood in 1 days
* Subjects who have participated in another clinical trial within 28 days prior to the study start

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-06; Primary Completion 2002-08 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability between Ranbaxy and Schering (Claritin-D® 24 hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Saint-Laurent, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html